CLINICAL TRIAL: NCT02257333
Title: High Focused Evaluation of Atherosclerotic Risk Profile in Retinal Thrombosis: Vascular Events Incidence, Sex Involvement and Interventional Outcomes Assessed by Ophthalmologists and Internists Network
Brief Title: Retinal Thrombosis and Atherosclerosis
Acronym: HEART-VISION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Stefania Basili, Associate Professor, University of Roma La Sapienza
Other Study IDs: HEART VISION
Record Dates: First submitted 2014-09-26; First posted 2014-10-06 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Retinal Vein Occlusion
Keywords: Retinal Vein Occlusion; Atherosclerosis; Risk Factors; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Retinal Vein Occlusion; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The retinal vein occlusion (RVO) is the second most common retinal disease after diabetic retinopathy, and is a common cause of unilateral visual loss. The risk factors that predispose to RVO are many and are generally the same as those found in vascular alterations involving other parts of the body, as in the case of stroke or coronary heart disease. Several authors have attempted to determine whether the pathogenesis of RVO can be of arterial type, considering the disease as consequent to atherosclerosis, rather than resulting from venous disease. Although less frequent than the other diseases RVO affects considerably on health care costs. Direct medical costs showed that in one year a patient with this disease has a higher than average cost for a patient with hypertension or glaucoma. Knowing the prevalence of the disease in Italy and identify modifiable risk factors, recognizing additional risk factors related to gender, genetic predisposition and especially the social-economic and cultural background in the pathogenesis of RVO, are the objectives that led to the planning of this study. In order to assess the prevalence of the disease and the current "clinical practice" we aim to create an online register between Italian specialist centers (ophthalmic emergency care and thrombosis centers) with immediate portability and usability of the data.

DETAILED DESCRIPTION:
The retinal vein occlusion (RVO) is the second most common retinal disease after diabetic retinopathy, and is a common cause of unilateral visual loss. The occlusion of a branch of the central retinal vein (BRVO) and central retinal vein occlusion (CRVO) are two topics discussed and very deserving of further study, especially for the need of greater clarity arising from the availability of new diagnostic and especially therapeutic opportunities.

The literature on the prevalence of RVO is not particularly rich, and the results of the available studies are very heterogeneous because such studies are conducted on a few cases, using different methodologies and are mainly characterized by a different distribution of risk factors among the different populations. In this regard, it was particularly interesting a publication of 2010 which proposed a combined analysis of the main study population (population based study).

The sample of the final analysis was of 49 869 subjects, and the results showed that the retinal vein occlusion overall prevalence, standardized for age and sex, is 5.2 per 1000, of which 4.42 and 0.80 to BRVO and CRVO respectively. Despite the slightly higher prevalence in females, this difference wasn't statistically significant.

In contrast, the prevalence of venous occlusion increases with increasing age in a statistically significant manner, both in the overall analysis of the occlusions of branch and central, that for the individual entities. This pattern is characteristic of chronic degenerative diseases and in fact the RVO has a behavior very similar to that of these diseases, probably because the risk factors (especially those such as atherosclerosis and systemic hypertension) increases with age.

The results provided by these systematic analysis are particularly important because they provide a reliable estimate of RVO prevalence in general population; must be considered, however, the inherent limitations mainly concerning potential sources of heterogeneity, such as different methodologies used, the fact that most of the studies were carried out on a single ethnic group, often with different distribution of risk factors and therefore were not suitable to capture these differences.

The risk factors predisposing to RVO are many and are generally the same as those found in vascular alterations involving other parts of the body as in the case of stroke or coronary heart disease. Several authors have attempted to determine whether the disease can be consequent to atherosclerosis and therefore caused by arterial disease rather than the pathogenesis of venous disease.

There is a very variable delay between the onset of symptoms and initiation of treatment; the excessive delay of treatment was considered an exclusion criterion in only a minority of the studies considered. Although it is very difficult to estimate the age of the thrombotic event, early identification is surely preferable and the treatment time is a critical factor to evaluate the efficacy of a therapeutic strategy. Because of the relatively small number of patients is not possible to determine which therapy is more effective.

Recently new experimental therapeutic approaches have been proposed, such as intravitreal administration of various drugs (steroids, anti-VEGF). It is not yet clear whether these approaches can eliminate the need for anticoagulant therapy during the acute phase of the disease. Surely antithrombotic drugs may have a role in the treatment of the acute phase of the RVO, at least in some categories of patients, and can be used in association with intravitreal drugs. Future studies should also explore the possibility of combined approaches. The retinal vein occlusion is a disease related to age and surely there will be an increase in social-economic impact of this disease due to the increase in population of the most advanced age group.

To assess the social-economic impact should be considered in addition to visual impairment related to the disease, the impact on quality of life of the patient and the direct medical costs of retinal vein thrombosis have shown that in one year a patient with this disease has an average cost 20% higher than a hypertensive patient (BRVO: + 16%; CRVO: + 22%) or glaucoma ones (BRVO: + 18%; CRVO: + 24%); Therefore, although it is less frequent than the other diseases RVO affects considerably on health care costs. The data available in the literature show that in the overall one year management, direct costs that have the greatest impact, in percentage terms, are the costs associated with ocular pathology caused by acute event (thrombosis) and diagnostic tests. After three years, however, the cost is linked to systemic disease (hospitalization) has a bigger impact in percentage terms, as if to indicate that retinal vein thrombosis is nothing more than an epiphenomenon of systemic disease.

Operating Modes The study will be divided into 4 phases: Step 1: establishment of the network: identification of specialized facilities (ophthalmic emergency care and thrombosis centers), which may accept patients with suspected RVO, which will participate in the establishment of the register online; Step 2: Create the registry and recruitment of patients cohort; Step 3: Follow-up planned (1 month) for instrumental tests to confirm the diagnosis of RVO; Step 4: Observational follow-up supported by dedicated web platform for the identification of major adverse cardiovascular events, in order to export in the context of clinical acquisitions epidemiological and disease management in real time.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Suspicion of Retinal Vein Occlusion
* Written Informed Consent

Exclusion Criteria:

* Pregnancy
* Short Life Expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with clinical suspicion of Retinal Venous Occlusion, consecutively enrolled at specialized ophthalmologic centers afferent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Retinal Venous Occlusion Prevalence | Baseline
  The primary outcome result is about the description of RVO prevalence among the study population.

SECONDARY OUTCOMES:
Atherosclerotic Risk Profile in RVO | Baseline
  The second primary outcome is to identify and describe the atherosclerotic burden and the atherosclerosis risk factors prevalence among RVO patients.
Visual Acuity | 2 Years
  To evaluate visual acuty in a long time frame after RVO. Visual acuity will be assessed according to Snellen and ETDRS scales.
Major Adverse Cardiovascular Events | 2 Years
  Evaluate incidence and prevalence of MACE among patients with RVO
RVO Recurrence | 2 Years
  It will be evaluated wheter the first RVO episode could be a risk factor for the occurence of a new RVO.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Basili, MD, Study Chair — University of Roma La Sapienza; Elena Pacella, MD, Study Chair — University of Roma La Sapienza; Enzo M Vingolo, MD, Principal Investigator — University of Roma La Sapienza; Valeria Raparelli, MD, PhD, Principal Investigator — University of Roma La Sapienza; Marco Proietti, MD, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome - Policlinico Umberto I Roma, Rome, I, Italy